CLINICAL TRIAL: NCT03646045
Title: Transpyloric Feeding for Prevention of Micro-aspiration
Status: Active, not recruiting | Type: Observational
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Zubair Aghai, Professor of Pediatrics, Nemours Children's Clinic
Other Study IDs: 741563-9
Record Dates: First submitted 2018-07-30; First posted 2018-08-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Microaspiration; Gastro Esophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tracheal aspirate samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transpyloric feed: Preterm infant receiving transpyloric feeding.
  Interventions: Other: Transpyloric feeding
- Control: Preterm infants receiving gastric feeding

INTERVENTIONS:
Other: Transpyloric feeding — Preterm infant feeding using transpyloric feeding tube (nasoduodenal tube)
  Groups: Transpyloric feed

SUMMARY:
To determine the effect of transpyloric (TP) feeding on microaspiration and lung inflammation in ventilated preterm infants.

DETAILED DESCRIPTION:
Specific Aim 1): To determine the effect of TP feeding on microaspiration and lung inflammation. Hypothesis: TP feeding will reduce the microaspiration and pulmonary inflammation in ventilated preterm infants. Evaluate markers of microaspiration (pepsin A) and lung inflammation [total cell counts, nuclear factor-kB (NF-kB) activation, tumor necrosis factor-α (TNF-α), IL-1β, IL-6, IL-8, angiopoietin 2 (Ang2), high-mobility group box-1 protein (HMGB1), macrophage migration inhibitory factor (MIF) and interferon-γ (IFN-γ)] in TA samples obtained from preterm ventilated infants with and without TP feeding.

Specific Aim 2): To determine the effect of TP feeding on respiratory support. Hypothesis: TP feeding will decrease the respiratory severity score (RSS) [Fraction of inspired oxygen (FiO2) X mean airway pressure (MAP)] and number of infants requiring ventilator support. Evaluate respiratory support in preterm ventilated infants with and without TP feeding.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with birth weight <1500 grams
* Requiring ventilatory support

Exclusion Criteria:

* Culture-proven sepsis
* Ventilator associated pneumonia (VAP).

Ages: 0 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants (birth weight <1500 grams) requiring ventilator support.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2016-11-04 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Tracheal aspirate pepsin A levels in ventilated preterm infants receiving transpyloric feeding and gastric feeding. | 3-7 days
  Difference in tracheal aspirate pepsin A levels in preterm ventilated infants receiving transpyloric feeding and gastric feeding.

SECONDARY OUTCOMES:
Tracheal aspirate pepsin A levels in ventilated preterm infants before and after transpyloric feeding. | 3-7 days
  Change in tracheal aspirate pepsin A levels in preterm ventilated infants before and after transpyloric feeding.
Tracheal aspirate cytokines levels (TNF-α, IL-1β, IL-6, IL-8, Ang2, HMGB1, MIF and IFN-gamma) in ventilated preterm infants receiving transpyloric feeding and gastric feeding. | 3-7 days.
  Difference in tracheal aspirate cytokines levels (TNF-α, IL-1β, IL-6, IL-8, Ang2, HMGB1, MIF and IFN-gamma) in preterm ventilated infants receiving transpyloric feeding and gastric feeding.
Tracheal aspirate cytokines levels (TNF-α, IL-1β, IL-6, IL-8, Ang2, HMGB1, MIF and IFN-gamma) in ventilated preterm infants before and after transpyloric feeding. | 3-7 days
  Change in tracheal aspirate cytokines levels (TNF-α, IL-1β, IL-6, IL-8, Ang2, HMGB1, MIF and IFN-gamma) in preterm ventilated infants before and after transpyloric feeding.
Respiratory support in ventilated preterm infants receiving transpyloric feeding and gastric feeding. | 7-14 days
  Difference in respiratory severity score (FiO2 X mean airway pressure) in preterm ventilated infants receiving transpyloric feeding and gastric feeding.
Respiratory support in ventilated preterm infants before and transpyloric feeding. | 7-14 days
  Change in respiratory severity score (FiO2 X mean airway pressure) in preterm ventilated infants before and after transpyloric feeding.

CONTACTS AND LOCATIONS:
Overall Officials: Zubair H Aghai, MD, Principal Investigator — Nemours
Locations (2):
- United States (2):
  - AI duPont Hospital for Children, Wilmington, Delaware
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No